CLINICAL TRIAL: NCT01570673
Title: Group Versus Individual Urotehrapy in Children With Non-neurogenic Lower Urinary Tract Dysfunction
Brief Title: Group Versus Individual Urotherapy for Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-089
Record Dates: First submitted 2012-04-02; First posted 2012-04-04 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2015-06

CONDITIONS: Lower Urinary Tract Symptoms
Keywords: quality of life; urinary bladder; symptoms; children
MeSH Terms: conditions — Lower Urinary Tract Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group Urotherapy (Experimental): Children in this arm wil receive group urotherapy in small groups with other children.
  Interventions: Behavioral: Group urotherapy
- Individual urotherapy (Active Comparator): Children will receive standard individual urotherapy in regular pediatric urology clinic.
  Interventions: Behavioral: Individual Urotherapy

INTERVENTIONS:
Behavioral: Group urotherapy — Children in this arm will receive group urotherapy in small groups with other children.
  Arms: Group Urotherapy
Behavioral: Individual Urotherapy — Children will receive standard individual urotherapy in regular pediatric urology clinic.
  Arms: Individual urotherapy

SUMMARY:
What are we doing? A pilot research study is planned to take place within the Pediatric Urology program at McMaster Children's hospital starting this spring/summer 2012. The pilot study will compare standard individual teaching that occurs in pediatric urology clinic about bladder re-training and achieving healthy bladder and bowel habits to a group teaching session. The group teaching session will be one hour in length and include the same content taught in pediatric urology clinic and provide more time for the children to ask questions, demonstrate and practice different exercises and talk about some of the challenges associated with having problems with their bladder. The group teaching session will be approximately one hour in length and occur weekly in the evenings for 12 to 15 weeks. Study participants will be asked to attend either one group teaching session or one individual teaching session which will occur in regular pediatric urology clinic. Parents will be asked to complete a demographics questionnaire at the start of the study and child participants will be asked to complete 2 short questionnaires about symptoms and quality of life before and after either individual or group teaching sessions. At the 3 month follow up, parents and child participants will also be asked to fill out an evaluation form of the session received. Children between the ages of 6 and 10 years old and a diagnosis of nonneurogenic lower urinary tract dysfunction will be asked if they would like to participate.

Why are we doing it? Some of the symptoms of bladder dysfunction include incontinence (wetting), recurrent urinary tract infections, frequency (having to pee a lot) and urgency (having sudden urges to pee). These symptoms can affect a child's physical and emotional/mental well-being. Treatment includes improving bladder habits through bladder re-training and improving bowel habits through treatment and management of constipation as well as establishing a bowel routine. Children are taught about their urinary tract system and what they need to do to improve and maintain its health. Children are asked to void (pee) every 2 hours, double void and drink more water. Sometimes they also need to take medications. Often in a busy clinic, parents are taught what the child needs to do and expected to return home and implement the bladder re-training instructions. Participation of the child during these visits varies. However, participation and engagement of the child in bladder re-training is crucial for success. Also, little time is spent on the impact of bladder dysfunction on the lives of these children. Many children do not want to follow the instructions on bladder re-training because they are worried about what their peers may say.

What do we hope to accomplish? The purpose of this study is to assess the feasibility of a group teaching session and evaluate the preliminary effectiveness of the session. Questionnaire results will be compared before and after the teaching sessions and between the individual and group teaching groups. Evaluation forms will provide feedback about the teaching sessions which will help determine the strengths of the sessions and improvements that could be made to improve the quality and effectiveness of future treatment. Outcomes that will be measured include symptoms and quality of life. This pilot study will also provide important information related to symptoms and quality of life for these children.

DETAILED DESCRIPTION:
Background Urotherapy has been the standard nonsurgical, nonpharmacologic treatment for children with nonneurogenic lower urinary tract dysfunction (NLUTD) and dysfunctional elimination syndrome (DES) for over two decades (Hoebeke, 2006). Children with NLUTD/DES represent a heterogenous group whose physical and mental health are affected (Afshar et al., 2009). There is no widely accepted diagnostic criteria (Afshar et al.) and urotherapy modalities that have been studied vary by setting, curriculum, length of treatment, outcome measurements and study participants. It is challenging to determine what modality of urotherapy is the most effective by reviewing the current literature. Furthermore, quality of life as an outcome measurement of urotherapy has not been reported in the literature.

Purpose The purpose of this study is to assess the feasibility of a group urotherapy session and evaluate the preliminary effectiveness of the group urotherapy session by measuring NLUTD/DES symptoms and quality of life and compare the group urotherapy session to standard urotherapy that takes place in pediatric urology clinics.

Methods Children aged 6-10 years old diagnosed with NLUTD/DES will be recruited from pediatric urology clinic at McMaster Children's Hospital over 12 to 15 weeks. The aim is to recruit at least 60 participants, 30 will be randomized to the control group and receive standard individual urotherapy in clinic and 30 will be randomized to the experimental group and receive a 1 hour group urotherapy session. Parents will be asked to complete a demographics questionnaire at the time of consent and children will be asked to complete 2 questionnaires at time of consent and again 3 months after receiving either individual or group urotherapy. At the 3 month follow up, parents and participants will be asked to complete an evaluation form to provide feedback about the teaching session received.

Outcome Measurements NLUTD/DES symptoms will be evaluated using the Vancouver NLUTD/DES questionnaire. This questionnaire assesses the following symptoms: incontinence, urgency, frequency, dysuria, hesitancy, straining and constipation. Quality of life (QOL) will be measured using the PinQ QOL measure. This questionnaire measures 6 domains of QOL: social, self-esteem, family, body image, independence and mental health. Both questionnaires have been deemed valid and reliable in children with the same diagnosis and age as the study population.

Impact This pilot study will provide new knowledge as a controlled trial comparing standard individual and group urotherapy which has not been reported on in the literature. Urotherapy is effective, but the search for the most effective program continues. This pilot study will provide information on the feasibility of the group urotherapy session as well as preliminary effectiveness. Furthermore, quality of life as an outcome measure has not been used to evaluate urotherapy. Again, this will provide new and valuable knowledge on the child's perception of their condition and the effect of urotherapy on their QOL.

References Afshar, K., Mirbagheri, A., Scott, H. & MacNeily, A.E. (2009). Development of a syndrome score for dysfunctional elimination syndrome. The Journal of Urology, 182, 1939-1944.

Bower, W.F., Sit, F.K.Y., Bluyssen, N., Wong, E.M.C. & Yeung, C.K. (2006). PinQ: A valid, reliable and reproducible quality-of-life measure in children with bladder dysfunction. Journal of Pediatric Urology, 2, 185-189.

Hoebeke, P. (2006). Twenty years of urotherapy in children: what have we learned? European Urology,49, 426-428.

ELIGIBILITY:
Inclusion Criteria:

* children aged 6-10 years of age with a diagnosis of NLUTD or DES based on history and physical examination.

Exclusion Criteria:

* grade 3 or 4 hydronephrosis; grade 3, 4, 5 vesicoureteral reflux; other diagnosis which affects bladder/bowel function (i.e. Spina Bifida); English as a second language; diagnosed learning disability (i.e. Attention Deficit Disorder, Attention Deficit Hyperactivity Disorder), mental health condition (i.e. anxiety, depression) and cannot have received urotherapy within the past 24 months.

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2012-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
lower urinary tract symptoms | 3 months
  incontinence, urgency, frequency, dysuria, hesitancy, straining and constipation

SECONDARY OUTCOMES:
quality of life | 3 months
  quality of life related to bladder/bowel health

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster Children's Hospital, Hamilton, Ontario, Canada